CLINICAL TRIAL: NCT00954148
Title: Defining the Utility of PET/CT in the Follow-up of Patients With Solid Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1st years Enrollment #s showed study was not going to meet criteria randomization.
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Thomas Anthony, MD Chief of Surgery, VANTXHCS Dallas, TX
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 09-017
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-05

CONDITIONS: Cancer Recurrence; Solid Tumors
Keywords: cancer; colorectal; head/neck; lung; PET/CT
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PET/CT follow-up (Active Comparator): PET/CT with history and physical exams at 3,9,18,36,60 months only
  Interventions: Procedure: PET/CT
- conventional follow-up (Other): NCCN recommendations
  Interventions: Procedure: NCCN recommendations for solid tumor post treatment

INTERVENTIONS:
Procedure: PET/CT — 5 visits with PET/CT as only testing
  Arms: PET/CT follow-up
Procedure: NCCN recommendations for solid tumor post treatment — 12-14 visits with exams, blood tests, CTs and PET/CT
  Arms: conventional follow-up

SUMMARY:
This is a comparison, at this VA Hospital,of routine multi-visit and multi-testing for solid tumor recurrence in four tumor groups to a limited scheduled 5 visit history/physical with PET/CT only, over a five year period. The purpose is to show through utilization of the single most sensitive and specific test currently available-PET/CT-that survival for patients in follow-up can be improved.(Plus lowering medical costs and increasing patient confidence and compliance with follow-up appointments).

DETAILED DESCRIPTION:
Routine visits would include COLON:14 visits with cea and 6 CTs over a 5 year period plus PET/CT at last visit RECTAL: 14 visits with cea and 6 CTs and 4 procto exams over 5 year period plus PET/CT at last visit HEAD/NECK: 14 visits with 4 CTs and PET/CT at last visit LUNG:12 visits plus 4 CTs and PET/CT at last visit

Limited follow-up ALL GROUPS: a history and physical plus PET/CT at 3 month, 9 month, 18 month, 36 month and 60 month only

ELIGIBILITY:
Inclusion Criteria:

* Completed primary therapy such that no disease is evident at the time of enrollment in the study

Exclusion Criteria:

* Patients unable to consent
* Without diagnosis of colorectal cancer
* Non-small cell lung cancer or squamous cell cancer of the head and neck
* Unwilling or unable to participate in the assigned follow-up program
* Having a serum glucose at time of PET/CT greater than 180mg/dl
* Stage IV disease or with evidence of disease recurrence post treatment
* Who are not a candidate for further treatment should a recurrence of disease be identified

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
ThatPET/CT will be superior (15% improvement) to conventional methods of follow-up in terms of 5 year survival, cost and time to identification of new disease | 5 years

SECONDARY OUTCOMES:
Improvement in patient/caregiver compliance in keeping their appointments and completing their tests | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: James LePage, PH.D, Study Chair — ACOS for Research VA North TX Health Care System
Locations (1):
- VA North Texas Health Care System, Dallas, Texas, United States